CLINICAL TRIAL: NCT03916848
Title: Novel Network Analysis of Intracranial Stereoelectroencephalography
Acronym: NNAIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18NM09
Record Dates: First submitted 2019-04-04; First posted 2019-04-16 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Epilepsy in Children; Focal Epilepsy; Epilepsy Intractable; Epilepsy, Focal; Intractable Epilepsy; Refractory Epilepsy; Epilepsies, Partial
Keywords: Stereoelectroencephalography; Single unit recording; Single neuron recording; SEEG; Epilepsy surgery
MeSH Terms: conditions — Epilepsies, Partial; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined Micro-Macro SEEG Electrodes (Experimental): Implanting SEEG electrodes with combined micro-macro electrodes capable of recording clinical data and experimental micro electrode single unit data
  Interventions: Procedure: Combined Micro-Macro SEEG Electrodes

INTERVENTIONS:
Procedure: Combined Micro-Macro SEEG Electrodes — The novel combined micro-macro electrodes will then be used during the surgical implantation procedure. The use of these novel electrodes will not change the surgical procedure, which is conducted using robotic assistance to ensure optimal accuracy. The macro electrode recordings will be used for routine clinical analysis and the duration of recording and subsequent analysis of the recordings will not be affected by the micro electrode data captured for research purposes. The clinical SEEG also involves electrical stimulation of the brain which will not be affected by the study.

SUMMARY:
Epilepsy is a disorder of the brain which is associated with disabling seizures and affects 100,000 people under 25. Many children with epilepsy also have a learning disability or problems with development. Although better outcomes occur in children who are successfully treated early for their epilepsy, 25% continue to have seizures despite best medical treatment.

One potential treatment is a neurosurgical operation to remove parts of the brain that generate seizures. A proportion of these children have electrodes inserted into their brains as part of their clinical assessment, termed stereoelectroencephalography (SEEG), to help localise these regions. Subsequent surgery is not always successful - up to 40% of children will have ongoing seizures 5 years after surgery.

The purpose of this study is to assess the utility of specially designed SEEG electrodes which can measure signals from single brain cells. These electrodes record the same clinical information as normal SEEG electrodes and are implanted in the same way, but can give the research team extra information at the same time. The investigators aim to assess whether studying the changes in the firing of individual cells, both during and between seizures, improves our ability to localise seizures and therefore improve outcomes following surgery.

As part of this research project, the investigators will not be doing anything that is not already part of the normal investigation and treatment for these children. Children will be recruited to the study during routine outpatient clinic visits. Surgical planning and execution will not be affected. The electrodes are CE licensed for clinical use and do not alter the risks of the operation. Following the period of monitoring, the care of these children would not be altered in any way.

The investigators aim to recruit 30 patients over 3 years. In addition to dissemination via scientific publications and presentations, the findings will be shared with participants and the public.

DETAILED DESCRIPTION:
Hypothesis

The hypothesis is that analysis of ictal (during seizure) and interictal (between seizures) single neuronal firing dynamics will identify ictogenic tissue in children undergoing SEEG recording for focal epilepsy.

Study Design

Prospective cohort study.

Sample Size

The investigators will aim to recruit 30 patients over a period of 3 years, of which 50% will have a normal MRI and 50% will have an identifiable lesion. It is not possible to conduct specific sample size calculations for this study but the centre carries out approximately 24 SEEG recordings per year so this target is feasible and achievable.

Participant Journey

The current patient pathway for children with medically refractory epilepsy undergoing pre-surgical evaluation will not be altered by the current study. The suitability for SEEG recording will be determined by the specialist epilepsy multidisciplinary team (MDT) and patients and parents will be invited to the neurosurgical outpatient clinic to discuss the procedure. There is nothing additional that will be required as part of this research study.

If they agree to proceeding with the SEEG recording procedure, patients will be invited to participate in this study during routine outpatient clinic visits. The treating consultant neurosurgeon (who is part of the routine clinical care team) will inform the patients and parents about the study and give them the opportunity to meet with the clinical research fellow. Patients and their parents will have the study explained to them by the research fellow and be given age-specific information sheets. Following an adequate time to digest this information (a few weeks) and an opportunity to ask any questions, the child (if appropriate) and their parents will choose whether or not they wish to participate in the research. If they choose to participate they will be asked to give written informed consent.

The novel combined micro-macro electrodes will then be used during the surgical implantation procedure. The use of these novel electrodes will not change the surgical procedure, which is conducted using robotic assistance to ensure optimal accuracy. The macro electrode recordings will be used for routine clinical analysis and the duration of recording and subsequent analysis of the recordings will not be affected by the micro electrode data captured for research purposes. The clinical SEEG also involves electrical stimulation of the brain which will not be affected by the study. Participation in this study will not preclude participation in these other studies and it may be possible to use the micro electrode data to supplement analyses in these other studies. Subsequent decision making on suitability for a surgical procedure will follow the normal clinical pathway and will not be affected by the micro electrode recording data.

Further participant follow-up will be observational and data will be obtained from routinely available clinical information, including whether or not a surgical resection is carried out and, if so, whether the patient remains seizure-free at follow-up.

The pseudo-anonymised research data will be securely stored via a secure university (UCL) research data storage service in a safe haven. Data will be stored for the duration of the study and 15 years following completion of the study to comply with GOSH guidelines. Data will be analysed according to the pre-specified data analysis plan, outlined elsewhere in this application.

Timeline

* February 2019 - April 2019 (3 months): Study and infrastructure set-up including acquisition of appropriate recording amplifiers and finalisation of data storage arrangements.
* May 2019 - July 2021 (2 years 3 months): Recruitment. Aim to recruit 15 patients per year. Sufficient provision to allow for slow recruitment in the timeline to ensure that adequate sample is achieved for subsequent analysis.
* August 2021 - October 2021 (3 months): Data analysis.
* November 2021 - January 2022 (3 months): Write-up and dissemination of results. The scientific results will be disseminated in the form of peer-reviewed publications & conference presentations. In addition, sessions will be held to disseminate the results to patients and the public, in the form of information evenings to groups such as Young Epilepsy and Epilepsy Action.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing SEEG recording as part of the investigation of their epilepsy at Great Ormond Street Hospital for Children
* Aged 3-18
* Participant/parents provide informed consent for inclusion

Exclusion Criteria:

* Lack of informed consent

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Analyse single unit behaviour in different brain regions. | Recording will continue for a period of 5-10 days, as determined by the clinical team. We will therefore use the data collected over the entire recording period for analysis.
  We will assess the abnormalities in single neuron firing behaviour both during and between seizures in children undergoing stereoelectroencephalogaphy (SEEG) as part of work-up for epilepsy surgery.
  The statistical analysis will include measures of timing coding and population coding of these single units and the investigators will assess these properties in time periods both during and between seizures to assess whether neurons in the seizure onset zone behave differently to those outside the seizure onset zone:
  1. Timing coding is evaluated using a generalized linear modeling (GLM) approach. An output of the GLM is called a post-spike filter (PSF), which models the propensity for the same neuron to fire again over the course of the subsequent 0.7 seconds.
  2. Population coding is also evaluated using a GLM by calculating coupling filters (the amount of up and down regulation of all other recorded neurons given that an individual neuron has just fired).
Correlate firing activity of single units to the clinically defined seizure onset zone (SOZ) | Recording will continue for a period of 5-10 days, as determined by the clinical team. We will therefore use the data collected over the entire recording period for analysis.
  Currently, the seizure onset zone (SOZ) is determined by visual analysis of the SEEG recordings at the end of the monitoring period.
  We aim to compare the differences in single unit behaviour (as defined above) between and during seizures in neurons inside and outside this clinically defined SOZ to assess if there is a unique behaviour to these neurons.

CONTACTS AND LOCATIONS:
Overall Officials: Rod Scott, PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Currently no provision for IPD sharing, will need further ethical approvals to do this.